CLINICAL TRIAL: NCT04057352
Title: The Citadel Embolization Device Study
Brief Title: Citadel Embolization Device Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDM10001448
Record Dates: First submitted 2019-08-01; First posted 2019-08-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Unruptured Wide-neck Aneurysms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Citadel Embolization Device (Other): The Citadel Embolization Device is intended to endovascularly obstruct or occlude blood flow in intracranial aneurysms.
  Interventions: Device: Citadel Embolization Device

INTERVENTIONS:
Device: Citadel Embolization Device — The Citadel Embolization Device is intended to endovascularly obstruct or occlude blood flow in intracranial aneurysms.

SUMMARY:
The purpose of this study is to gather safety and effectiveness data on Stryker Neurovascular's Next Generation Target Detachable Coil (hereafter referred to as the Citadel Embolization Device), when used with Target Detachable Coils, in the treatment of wide-neck intracranial aneurysms.

DETAILED DESCRIPTION:
In this study, use of the Citadel Embolization Device will be limited to a population of patients with unruptured or ruptured wide-neck aneurysms who meet all study eligibility criteria. The Citadel Embolization Device is intended to endovascularly obstruct or occlude blood flow in intracranial aneurysms.

ELIGIBILITY:
Inclusion Criteria:

1. Age is ≥18 and ≤80 years
2. Has a single, unruptured or ruptured target intracranial aneurysm that is suitable for endovascular treatment. Definition: For the purposes of this study, a ruptured intracranial aneurysm is defined as one with CT/MRI/LP evidence of subarachnoid hemorrhage attributed to the index aneurysm within the last 60 days.
3. Aneurysm morphology is saccular
4. Aneurysm size is between 6-12 mm
5. Has a wide-neck, saccular aneurysm, either bifurcation or sidewall, with a dome to neck ratio <2 or neck ≥4 mm
6. If the target intracranial aneurysm is classified as ruptured, patient must be neurologically stable with a Hunt & Hess Score of 1 or 2.
7. Must be willing to comply with protocol required procedures and follow up
8. Subject or LAR must be willing to sign and date an IRB approved written informed consent prior to initiation of any screening or study procedures

Exclusion Criteria:

1. Target aneurysm has been previously treated
2. Target aneurysm is in any extradural location, including the extradural cavernous segment
3. Has vessel characteristics, tortuosity or morphology or unfavorable aneurysm morphology (e.g., determined from baseline or preprocedure imaging, or which may be evidenced by excessive resistance felt during the procedure) that would preclude safe endovascular access to the target aneurysm necessary for treatment with the study device
4. Has significant intracranial atherosclerotic disease or stenosis determined from baseline or pre-procedure imaging
5. If the target intracranial aneurysm is classified as ruptured, patient is neurologically unstable or has a Hunt & Hess Score of ≥ 3
6. Has a history of intracranial vasospasm not responsive to medical therapy
7. Has undergone coiling or stenting of a non-target intracranial aneurysm within 30 days prior to study treatment or has a non-target intracranial aneurysm that is expected to be treated within 12 months following the treatment of the target aneurysm
8. Treatment with flow diverting stent implant is anticipated
9. A planned, staged procedure is anticipated
10. Has Moya-Moya disease, arteriovenous malformation(s), arteriovenous fistula(e), intracranial tumor(s), intracranial hematoma(s), any other intracranial vascular malformation, or any previous major intracranial surgery
11. Has had a recent (within 90 days) ischemic stroke, TIA, or intracranial hemorrhage
12. Has a baseline mRS score ≥2
13. Has a known coagulopathy or is on chronic anticoagulant therapy
14. Is pregnant or intends to become pregnant during the study or is breastfeeding
15. Is concurrently involved in another study that could affect outcomes of IA treatment
16. Has evidence of active cancer, terminal illness, high risk of embolic stroke, unstable atrial fibrillation, significant co-morbidities, major surgery ≤ 30 days pre-procedure, psychiatric disorders, substance abuse, or a life expectancy of less than 5 years
17. Has a contraindication to angiography, radiographic contrast agents, or any medications that are typically used during the procedure, and any other contraindications listed in the Investigational DFU
18. Has a confirmed allergy to platinum, tungsten, nickel (e.g. nitinol), or other elements used in the manufacturing of the investigational device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint is stroke-related neurologic death, or major ipsilateral or disabling stroke in the territory supplied by the treated artery | 12 months post-procedure
  Occurring within 12 months post-procedure as adjudicated by an independent Clinical Events Committee (CEC)
  * With major ipsilateral stroke defined as a stroke associated with an increase in NIHSS score ≥ 4 points persisting ≥ 24 hours, and;
  * With disabling stroke defined as a stroke that results in a modified Rankin Scale (mRS) score ≥ 3 assessed at a minimum of 90 days post-stroke event.
Primary Effectiveness Endpoint of this study is adequate aneurysm occlusion without retreatment or significant parent artery stenosis (>50% stenosis). | 12 months post-procedure
  The determination of adequate aneurysm occlusion using Raymond-Roy classification will be made if either of the following criteria in the description are met:
  -100% occlusion (Raymond Class I) demonstrated by Digital Subtraction Angiography (DSA) measurement at 12 months (± 3 months) post-procedure, or -Stable Raymond class II demonstrated on 2 serial imaging measurements using Contrast-Enhanced Magnetic Resonance Angiography (CE-MRA) and/or DSA obtained a minimum of 6 months (± 1 month) apart. Post-procedure and 12-month imaging must be completed with DSA.

SECONDARY OUTCOMES:
Secondary Safety Endpoint of this study is any stroke event occurring through 12 months post-procedure, where a stroke event is defined as per what is noted in the description. | 12 months post-procedure
  -Rapidly developing clinical signs of focal (or global) disturbance of cerebral function lasting more than 24 hours with no apparent cause other than of vascular origin, including ischemic stroke and/or hemorrhagic stroke (i.e., intraparenchymal hemorrhage [IPH], subarachnoid hemorrhage [SAH], subdural hemorrhage [SDH], epidural hemorrhage [EDH]) accompanied with radiological evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Ansaar Rai, MD, Principal Investigator — West Virginia University
Locations (26):
- United States (26):
  - Carondelet St. Joseph Hospital, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - California Pacific Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - John Muir Health, Walnut Creek, California
  - RIA Neurovascular, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - Baptist Health, Jacksonville, Florida
  - University of Miami/Jackson Memorial, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Indiana Methodist, Indianapolis, Indiana
  - Kansas University Medical Center, Kansas City, Kansas
  - Baptist Health, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - UMass Memorial Health, Worcester, Massachusetts
  - McLaren Health Center, Flint, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Washington University, St Louis, Missouri
  - Weill Cornell, New York, New York
  - Montefiore Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Washington, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No